CLINICAL TRIAL: NCT03273907
Title: Post Approval Study of the CyPass System in Patients With Primary Open Angle Glaucoma Undergoing Cataract Surgery
Brief Title: Post Approval Study of the CyPass System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Voluntary market withdrawal
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLD122c-C001
Record Dates: First submitted 2017-09-05; First posted 2017-09-06 (Actual); Results first posted 2022-09-21 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2022-08

CONDITIONS: Primary Open-angle Glaucoma; Cataract
Keywords: CyPass Micro-Stent
MeSH Terms: conditions — Glaucoma, Open-Angle; Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CyPass System (Experimental): CyPass Micro-Stent implanted with CyPass 241-S applier in the angle of the eye during cataract surgery
  Interventions: Device: CyPass Micro-Stent implanted with CyPass 241-S applier; Procedure: Cataract surgery

INTERVENTIONS:
Device: CyPass Micro-Stent implanted with CyPass 241-S applier — CyPass System (Model 241-S) consists of the CyPass Micro-Stent contained in a loading device (loader) and the CyPass applier.The CyPass Micro-Stent is an implantable medical device intended for long term use.
Procedure: Cataract surgery — Cataract surgery, followed by implantation of the CyPass Micro-Stent in one eye (the study eye) at the surgery visit

SUMMARY:
The purpose of this study is to demonstrate that the rate of clinically relevant complications associated with CyPass Micro-Stent placement and stability using the CyPass 241-S applier, as determined at 36 months in the postmarket setting, is less than the pre-specified performance target, which is based on experience with the CyPass Model E applier in COMPASS trial TMI-09-01 (NCT01085357).

DETAILED DESCRIPTION:
Each subject's expected participation in the study is up to 37.5 months which includes up to 42 days between the screening and surgery visits, and 36 months of post-surgery follow-up. Only one eye per subject will be implanted.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the requirements of the study and willing to follow study instructions, provide written informed consent, and agree to comply with all study requirements, including the required study follow-up visits
* Diagnosis of primary open angle glaucoma (POAG)
* Medicated intraocular pressure (IOP) of ≥10 millimeters mercury (mmHg) and ≤25 mmHg, or an unmedicated IOP of ≥21 mmHg and ≤33 mmHg
* An operable age-related cataract eligible for phacoemulsification
* Visual acuity as specified in the protocol
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Inability to complete a visual field test prior to surgery
* Use of ocular hypotensive medication/s, as specified in the protocol
* Diagnosis of glaucoma other than POAG, as specified in the protocol
* Other medical conditions, as specified in the protocol
* Proliferative diabetic retinopathy
* Previous surgery for retinal detachment
* Previous corneal surgery
* Wet age-related macular degeneration
* Poor vision in the non-study eye not due to cataract
* Significant ocular inflammation or infection within 30 days of screening visit
* Uncontrolled systemic diseases that may put the subject's health at risk and/or prevent the subject from completing all study visits
* Women who are pregnant or nursing
* Other protocol-specified exclusion criteria may apply.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Trial Lead, Surgical, Study Director — Alcon Research, LLC
Locations (20):
- United States (20):
  - Alcon Investigative Site, Phoenix, Arizona
  - Alcon Investigative Site, Orange, California
  - Alcon Investigative Site, Fort Collins, Colorado
  - Alcon Investigative Site, Jacksonville, Florida
  - Alcon Investigative Site, Panama City, Florida
  - Alcon Investigative Site, Gainesville, Georgia
  - Alcon Investigative Site, Marietta, Georgia
  - Alcon Investigative Site, Garden City, Kansas
  - Alcon Investigative Site, Fraser, Michigan
  - Alcon Investigative Site, St Louis, Missouri
  - Alcon Investivative Site, St Louis, Missouri
  - Alcon Investigative Site, Vineland, New Jersey
  - Alcon Investigative Site, Bala-Cynwyd, Pennsylvania
  - Alcon Investigative Site, Chambersburg, Pennsylvania
  - Alcon Investigative Site, Austin, Texas
  - Alcon Investigative Site, El Paso, Texas
  - Alcon Investigative Site, Houston, Texas
  - Alcon Investigative Site, Bellevue, Washington
  - Alcon Investigative Site, Kenosha, Wisconsin
  - Alcon Investigative Site, Racine, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 20 investigative sites located in the United States.
  Due to the CyPass voluntary global market withdrawal, enrollment was permanently suspended for this study starting 29 August 2018.
Pre-assignment Details: Of the 79 enrolled, 36 subjects were exited from the study prior to attempted implantation with the CyPass Micro-Stent. This reporting group includes all subjects with attempted implantation (43). Only one eye per subject was implanted.
Period: Overall Study
Arm/Group | CyPass System
Started | 43
Completed | 34
Not Completed | 9
Not completed — Death | 1
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 2
Not completed — COVID 19 | 2

BASELINE CHARACTERISTICS:
Population: Intent to Treat Analysis Set: All study eyes for which a CyPass Micro-Stent implant was attempted
Arm/Group | CyPass System
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.4 (5.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 41
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 35
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With Clinically Relevant Complications Associated With CyPass Micro-Stent Placement and Stability as Determined at Month 36
Description: Device-related complications, as specified in the protocol, included:
  * Failure to implant CyPass, defined as inability to successfully deploy or insert the CyPass.
  * Clinically significant CyPass malposition, defined as CyPass positioning after deployment such that:
    * The device is not in the supraciliary space, or
    * Clinical sequela resulting from device position including, but not limited to:
      * Secondary surgical intervention to modify device position (eg, repositioning, proximal end trimming or explantation)
      * Corneal endothelial touch by device
      * Corneal edema leading to loss of BCDVA > 2 lines at the last postoperative visit, in comparison with preoperative BCDVA
      * Progressive ECL, defined as ongoing reduction in endothelial cell count of 30% or more relative to the screening ECD value, where 'ongoing reduction in endothelial cell count' is defined as losses continuing after Visit 5 (6 Month Follow-up).
Time Frame: Up to Month 36 postoperative
Population: Intent-to-Treat (ITT) Analysis Set
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | CyPass System
Number analyzed (Participants) | 43
Number analyzed (eyes) | 43
percentage of eyes | 2.3
Statistical Analysis 1: Comparison: CyPass System; Test type: Superiority — The primary null hypothesis tested was that the observed rate of clinically relevant complications associated with CyPass Micro-Stent placement and stability is greater than or equal to the performance target rate of 7.00 percent; p = 0.1870, Exact one-sided binomial test; P-value is provided from exact one-sided binomial test with type I error 0.05 comparing CyPass System with performance criterion of 7.00 percent

2. Secondary Outcome: Mean Change in IOP From Baseline at Month 36
Description: Intraocular pressure (IOP) was assessed by Goldman tonometry and measured in millimeters mercury (mmHg). A negative change value indicates an improvement.
Time Frame: Baseline, Month 36 postoperative
Population: ITT Analysis Set with data at visit
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | CyPass System
Number analyzed (Participants) | 34
Number analyzed (eyes) | 34
mmHg | -3.71 (4.881)

3. Secondary Outcome: Percentage of Eyes With IOP Reduction 20 Percent or More From Baseline While Using the Same or Fewer Topical Ocular Hypotensive Medications at Month 36
Description: Intraocular pressure (IOP) was assessed by Goldman tonometry and measured in millimeters mercury (mmHg). A reduction in IOP from baseline indicates an improvement.
Time Frame: Baseline, Month 36 postoperative
Population: ITT Analysis Set with data at visit
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | CyPass System
Number analyzed (Participants) | 34
Number analyzed (eyes) | 34
percentage of eyes | 41.2 [24.6 to 59.3]

4. Secondary Outcome: Percentage of Eyes Not Using Ocular Hypotensive Medication With IOP ≥ 6 mmHg and ≤ 18 mmHg at Month 36
Description: Intraocular pressure (IOP) was assessed by Goldman tonometry and measured in millimeters mercury (mmHg). Only one eye per subject was implanted.
Time Frame: Month 36 postoperative
Population: ITT Analysis Set with data at visit
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | CyPass System
Number analyzed (Participants) | 34
Number analyzed (eyes) | 34
percentage of eyes | 61.8 [43.6 to 77.8]

5. Secondary Outcome: Percentage of Eyes With Sight-threatening Adverse Events (AEs)
Description: Sight-threatening adverse events, as specified in the protocol, included:
  * Persistent Best Corrected Distance Visual Acuity (BCDVA) loss of 3 lines or more
  * Endophthalmitis
  * Corneal decompensation
  * Retinal detachment
  * Severe choroidal hemorrhage or detachment
  * Aqueous misdirection. Note: If an eye had multiple occurrences of an AE, the eye is presented only once in the respective eye count column (n) for the corresponding AE.
Time Frame: Up to Month 36 postoperative
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | CyPass System
Number analyzed (Participants) | 43
Number analyzed (eyes) | 43
percentage of eyes | 2.3 [0.1 to 12.3]

6. Secondary Outcome: Percentage of Eyes With Ocular Secondary Surgical Interventions (SSI)
Description: A secondary surgical intervention may have occurred for any of the following reasons:
  * CyPass device explantation associated with CyPass placement and stability
  * CyPass device explantation NOT associated with CyPass placement and stability
  * Unplanned ocular surgical reintervention associated with CyPass placement and stability
  * Unplanned ocular surgical reintervention NOT associated with CyPass placement and stability (as defined in the protocol).
  Note: If an eye had multiple occurrences of an AE, the eye is presented only once in the respective eye count column (n) for the corresponding AE
Time Frame: Up to Month 36 postoperative
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | CyPass System
Number analyzed (Participants) | 43
Number analyzed (eyes) | 43
percentage of eyes | 7.0 [1.5 to 19.1]

7. Secondary Outcome: Percentage of Eyes With Ocular SSIs Associated With CyPass Placement and Stability
Description: A secondary surgical intervention may have occurred for either of the following reasons:
  * CyPass device explantation associated with CyPass placement and stability
  * Unplanned ocular surgical reintervention associated with CyPass placement and stability.
  Note: If an eye had multiple occurrences of an AE, the eye is presented only once in the respective eye count column (n) for the corresponding AE
Time Frame: Up to Month 36 postoperative
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | CyPass System
Number analyzed (Participants) | 43
Number analyzed (eyes) | 43
percentage of eyes | 2.3 [0.1 to 12.3]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected pre-treatment (Day -42 to Day -1) up to Month 36 Follow-up/Exit (Day +1050 to Day 1140). AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator.
Description: This analysis population includes all study eyes for which a CyPass Micro-Stent implant was attempted (Intent to Treat Analysis Set). "At Risk" population of pre-treatment and systemic AEs is reported in units of subjects; ocular AE population is reported in units of eyes.
Groups:
- Pretreatment: Events reported in this group occurred prior to attempted implantation with the test article
- CyPass Study Eye: Events reported in this group occurred after attempted implantation with the test article and include ocular events in the study eye
- CyPass Systemic: Events reported in this group occurred after attempted implantation with the test article and include systemic adverse events plus ocular events in the non-study eye
Arm/Group | Pretreatment | CyPass Study Eye | CyPass Systemic
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/43 | 1/43
Serious Adverse Events (participants affected / at risk) | 0/43 | 4/43 | 7/43
Other Adverse Events (participants affected / at risk) | 3/43 | 13/43 | 21/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pretreatment (N=43) | CyPass Study Eye (N=43) | CyPass Systemic (N=43)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Intraocular pressure increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Paracentesis eye (Investigations) | 0 (0) | 2 (2) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Throat cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Visual field defect (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Glaucoma drainage device placement (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pretreatment (N=43) | CyPass Study Eye (N=43) | CyPass Systemic (N=43)
Posterior capsule opacification (Eye disorders) | 0 (0) | 6 (6) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 3 (3) | 0 (0)
Intraocular pressure increased (Investigations) | 0 (0) | 4 (4) | 3 (3)
Visual field defect (Nervous system disorders) | 0 (0) | 3 (4) | 1 (1)
Cataract operation (Surgical and medical procedures) | 3 (3) | 0 (0) | 19 (19)

LIMITATIONS AND CAVEATS:
Considering the achieved sample size in this study (less than 10% of intended), no definitive conclusion can be made with respect to the rate of CyPass-related complications.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2017-08-22): https://cdn.clinicaltrials.gov/large-docs/07/NCT03273907/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/07/NCT03273907/SAP_001.pdf